CLINICAL TRIAL: NCT05038293
Title: Efficacy of Plaque Removal of a Novel Brushing Device Compared to a Manual Toothbrush
Brief Title: Efficacy of Plaque Removal of a Novel Brushing Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Diane M Daubert RDH, MS, PhD, Clinical Associate Professor: School of Dentistry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00013154
Record Dates: First submitted 2021-07-22; First posted 2021-09-09 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Dental Plaque
Keywords: Gingivitis; toothbrushing; oral hygiene; biofilm
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Intervention Model Description: Single-blind, parallel group, randomized controlled clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes assessors and the principal investigator will be blind to toothbrush device assignment. In order to maintain blinding and eliminate assessor bias, study team members instructing and observing participants in the use of the assigned toothbrushing device will not be outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Automated mouthpiece-based toothbrush (Experimental): Under observation of study staff, participants assigned to the automated mouthpiece-based toothbrush will insert a properly fitted mouthpiece and use the automated device directly over the sink.
  Interventions: Device: Automated mouthpiece-based toothbrush
- Manual toothbrush (Active Comparator): Under observation of study staff, participants assigned to the manual toothbrush will be timed brushing their teeth directly over the sink using a pre-dispensed quantity of toothpaste on bristles dampened with water.
  Interventions: Device: Manual toothbrush

INTERVENTIONS:
Device: Automated mouthpiece-based toothbrush — One-time use during study visit.
  Other Names: Novel toothbrushing device
  Arms: Automated mouthpiece-based toothbrush
Device: Manual toothbrush — One-time use during study visit.
  Arms: Manual toothbrush

SUMMARY:
The purpose of this research study is to compare how a novel, automated mouthpiece-based toothbrushing device removes dental plaque compared to a manual toothbrush.

DETAILED DESCRIPTION:
Plaque is one of the main etiological factors in dental decay and the principal etiological factor for periodontal diseases. Although toothbrushes have greatly evolved, dexterity is still the key component to an efficient cleaning routine. The primary goal is to examine 60 participants to determine the efficacy of a new powered teeth cleaning device designed to bypass the variability of individual dexterity compared with manual toothbrushing.

This is a single-blind, randomized controlled trial. Sixty pediatric patients will be recruited for the study and randomized into treatment and control groups, subdivided into primary (20), mixed (20), and permanent dentition (20). Participants will be asked to abstain from brushing, flossing, gum or mouthwash use for 24 hours prior to the study visit. Plaque will be assessed using the Turesky Modification of the Quigley-Hein Plaque Index before and after a one-time brushing with the assigned study device. A soft tissue assessment will be conducted and intraoral photos taken pre- and post-brushing.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 5-17
* In good general health
* Fluent in English
* Parent or guardian willing and able to provide written informed consent
* Have 16 scorable teeth (non-crown/bridge/or full amalgams)
* Have had a dental cleaning and exam in the past 24 months

Exclusion Criteria:

* Advanced periodontal disease or severe gum disease
* Mouth or teeth pain that prevents brushing in any areas
* Intraoral piercings (tongue or lip) that cannot be removed
* Non-controlled diabetes
* Any autoimmune or infectious disease or any medical condition that would delay wound healing
* Untreated visible cavities or untreated dental work
* Oral or gum surgery in the previous 2 months
* Take antibiotic premedication for dental procedures
* Undergoing or require extensive dental or orthodontic treatment
* Current smoker
* Generalized recession over 1mm

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane M Daubert, RDH, MS, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, School of Dentistry, Regional Clinical Dental Research Center (RCDRC), Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited via flyers posted at the Center for Pediatric Dentistry at the University of Washington. If parents were interested they contacted the study coordinator for a phone screening.
Pre-assignment Details: 62 parents called for a phone screening. Of those,48 subjects presented for the first appointment but 6 were not enrolled due to not meeting inclusion and exclusion criteria. 42 subjects were consented and enrolled.
Period: Overall Study
Arm/Group | Automated Mouthpiece-based Toothbrush | Manual Toothbrush
Started | 24 | 18
Completed | 22 | 18
Not Completed | 2 | 0
Not completed — device was not operating properly for one subject. | 1 | 0
Not completed — one subject was dropped due to a behavioral issue | 1 | 0

BASELINE CHARACTERISTICS:
Population: 24 were enrolled but 2 dropped
Groups:
- Total: Total of all reporting groups
Arm/Group | Automated Mouthpiece-based Toothbrush | Manual Toothbrush | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 18 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — age, continuous
  years | 10.1 [5 to 17] | 10.8 [6 to 17] | 10.45 [5 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 18 | 17 | 35
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 22 | 18 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Dental Plaque Removal Efficacy Using Turesky Modification of the Quigley-Hein Plaque Index
Description: Average Change from baseline plaque index after brushing with the automated mouthpiece-based brushing device versus a manual toothbrush. The Turesky Modification of the Quigley-Hein Plaque Index evaluates 6 areas per tooth and gives a score from 0-5 with 0 being no plaque and 5 being the highest amount of plaque and the average score for all sites was used for analysis.
Time Frame: baseline,1 minute after brushing
Population: participants aged 5-17 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Automated Mouthpiece-based Toothbrush | Manual Toothbrush
Number analyzed (Participants) | 22 | 18
units on a scale | 0.29 [.287 to .293] | 0.6 [.578 to .628]

2. Secondary Outcome: Change From Baseline in Presence of Soft Tissue Abrasion After Use of Automated Mouthpiece-based Brushing Versus Manual Toothbrush
Description: Number of participants with soft tissue abrasion after brushing with the automated mouthpiece-based.brushing device versus a manual toothbrush. An intraoral soft tissue examination will be done before and after brushing and a binary scale will be used to note any areas of abrasion (yes or no). Outcome is the presence of any soft tissue abrasion that was not present prior to brushing.
Time Frame: baseline, 1 minute after brushing
Population: 5-17 year old subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Automated Mouthpiece-based Toothbrush | Manual Toothbrush
Number analyzed (Participants) | 22 | 18
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: baseline visit up to 1.5 hours. (study was one visit only)
Description: definition does not differ
Arm/Group | Automated Mouthpiece-based Toothbrush | Manual Toothbrush
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 2/22 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Automated Mouthpiece-based Toothbrush (N=22) | Manual Toothbrush (N=18)
minor abrasion (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — minor soft tissue abrasion from brushing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT05038293/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT05038293/SAP_001.pdf